CLINICAL TRIAL: NCT01700426
Title: Enhancing Treatment of Iron Deficiency and Iron Deficiency Anemia With an Antioxidant, Vitamin E
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-1234
Record Dates: First submitted 2012-09-21; First posted 2012-10-04 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-03

CONDITIONS: Iron Deficiency; Iron Deficiency Anemia
Keywords: Iron Deficiency; Iron Deficiency Anemia
MeSH Terms: conditions — Iron Deficiencies; Anemia, Iron-Deficiency | interventions — Vitamin E

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- iron (Active Comparator): Sixty-eight subjects found to have ID or IDA will be consented and randomized to one of the two treatment regimens (34 subjects per group). Liquid supplement preparations of iron (both groups), Vitamin E (test) and placebo (control) will be distributed by the research pharmacy at Children's Hospital Colorado.
  A commercial ferrous sulfate solution (Fer-In-Sol, 15 mg elemental Fe/mL; Mead Johnson, Inc, Evansville, IN) will be distributed to all qualifying participants for the study by the research pharmacy at Children's Hospital Colorado. The volume of the suspension will be individualized by the pharmacy to the infant's weight, to maintain consistent iron dosing at 6 mg/kg/day.
  Interventions: Drug: Vitamin E
- iron 2 (Active Comparator): Sixty-eight subjects found to have ID or IDA will be consented and randomized to one of the two treatment regimens (34 subjects per group). Liquid supplement preparations of iron (both groups), Vitamin E (test) and placebo (control) will be distributed by the research pharmacy at Children's Hospital Colorado.
  A commercial ferrous sulfate solution (Fer-In-Sol, 15 mg elemental Fe/mL; Mead Johnson, Inc, Evansville, IN) will be distributed to all qualifying participants for the study by the research pharmacy at Children's Hospital Colorado. The volume of the suspension will be individualized by the pharmacy to the infant's weight, to maintain consistent iron dosing at 6 mg/kg/day.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Vitamin E — A commercial Vitamin E preparation (Aqueous Vitamin E®, 15 IU/0.3 ml; SilaRx, Inc, Spring Valley, NY) will be used for the study, also on the recommendation of the Children's Hospital Colorado (CHC) research pharmacist. The Vitamin E dose will be 18 mg/day for all subjects randomized to the Vitamin E group.
  Other Names: Aqueous Vitamin E®, 15 IU/0.3 ml
  Arms: iron
Other: Placebo — The control group will receive an indistinguishable placebo preparation, which will be compounded by the CHC research pharmacy using the following inactive ingredients: purified water, polysorbate 80, sorbital, and propylene glycol. This suspension is stable for 6 months.
  Arms: iron 2

SUMMARY:
The study addresses treatment of iron deficiency, the most common nutritional deficiency that infants and young children encounter. With the knowledge that iron deficiency may irreversibly affect a baby's long-term neurodevelopment and behavior, the investigators are offering free screening blood draws at Children's Hospital Colorado to older babies and toddlers (9-24 months old). If their blood results indicate a serum ferritin of ≤ 15 micrograms/dL without the presence of an elevated C-reactive protein (CRP), they will be invited to continue in the intervention portion of the study, where they will receive iron supplements as well as vitamin E (or placebo) for an eight week treatment period. The rationale for the study is to test whether addition of Vitamin E, an antioxidant and anti-inflammatory agent, improves the treatment response to supplemental iron.

DETAILED DESCRIPTION:
Enhancing Treatment of Iron Deficiency and Iron Deficiency Anemia with an Antioxidant, Vitamin E

Synopsis/Abstract Iron Deficiency (ID) and Iron Deficiency Anemia (IDA) are common in older breastfed infants and toddlers. Treatment of 3-6 mg iron/kg/day is recommended by the American Academy of Pediatrics (AAP), but this regimen often results in only modest changes in iron status, despite being a substantially higher dose (relative to body weight) than is commonly used for adults. We propose that high therapeutic doses of iron induce an inflammatory response, thus increasing hepatic synthesis of a critical regulator of iron absorption, hepcidin, which functions to limit iron absorption in the context of inflammation. In infants and toddlers found to have ID or IDA, we propose to evaluate the efficacy of the addition of Vitamin E to iron therapy compared with the same dose of iron alone. Our primary hypothesis is that in infants and toddlers with ID or IDA, 2 months of supplemental Vitamin E combined with therapeutic iron supplementation will be more efficacious than the same dose of iron alone. The study design is a randomized, double blind efficacy trial of 2 months of iron therapy (6 mg/kg/day) with or without Vitamin E (18 mg/day), in infants and toddlers with ID or IDA from 9 to 24 months of age. Primary outcomes include biomarkers of iron status (ferritin, hemoglobin, transferrin saturation, and transferrin receptor); secondary outcomes include biomarkers of inflammation and oxidant stress. Subjects: We will screen older infants (9-12 months of age) who were predominantly breastfed through at least the first 9 months of life, and toddlers (12-24 months of age) who were breastfed and/or who have modest dietary iron intakes. Intervention: Sixty-eight subjects found to have ID or IDA will be consented and randomized to one of the two treatment regimens (34 subjects per group). Liquid supplement preparations of iron (both groups), Vitamin E (test) and placebo (control) will be distributed by the research pharmacy at The Children's Hospital.Children's Hospital Colorado. Outcomes: Biomarkers of iron status, iron homeostasis, oxidant stress, and of systemic and intestinal inflammation will be repeated at the end of the intervention. If the hypotheses are supported, the findings would provide a simple and effective modification to enhance iron therapy, and to improve the balance between adequate iron uptake to meet physiologic needs and excessive iron intake and its potential adverse effects.

I. Goals and objectives:

The broad goal of this proposal is to improve the health and nutrition of young children by improving iron status of infants and toddlers who have developed iron deficiency (ID) or iron deficiency anemia (IDA). The specific objective is to test an intervention proposed to enhance the efficacy, and minimize potential toxicity, of therapeutic iron for infants and young children who have a dietary iron deficiency.

Iron deficiency is the most common micronutrient deficiency in the world and negatively impacts health in several ways 1, 2. ID and IDA contribute to stunting and impaired growth, increased behavioral problems, and delayed mental and motor development 3, 4, 5-7. Studies have also shown that some of the behavioral and developmental consequences of ID and IDA in young children are not reversible with treatment 8. Despite the fortification of infant and toddler foods in the United States, a significant number of children still develop ID or IDA 9. Current treatment recommendations include a wide dosage range (3-6 mg/kg/day), which represents amounts that are higher than routine supplementation levels for adults (typically equivalent to < 1 mg/kg/day), reflecting the challenge and imprecision of effective treatment for ID and IDA in children. Iron excess is not without risk, and studies in adults have shown local (intestinal) and systemic inflammatory changes within days of iron therapy initiation 10, 11. Recent advances in the understanding of the regulation of iron homeostasis and metabolism indicate that systemic inflammation induces a protein called hepcidin, which blocks the uptake of iron into the body12, 13. Thus, stimulation of inflammation by high dose iron supplements may actually counteract the intended beneficial effect of the increase in iron intake.

Vitamin E is an essential nutrient that functions as an antioxidant and anti-inflammatory agent, and has been studied for many potentially beneficial facets of human health, including potential for protection against heart disease14; accelerated aging mediated through DNA damage; and impaired immunity 15. Research in adults giving antioxidants along with iron therapy was associated with reduced oxidative potential. In this study, a palm oil extract containing approximately 7 mg of Vitamin E was supplemented along with iron therapy and was associated with reduced fecal oxidation 16 Alpha-tocopherol is the most studied form of Vitamin E, and has been shown to decrease biomarkers of total body oxidative stress and inflammation 15, 17. We propose to accomplish our primary specific objective by testing the effect on treatment outcomes of administration of Vitamin E along with iron supplements.

II. Hypotheses:

Our central hypothesis is that in infants and toddlers with ID or IDA, 2 months of supplemental Vitamin E combined with therapeutic iron supplementation at 6 mg/kg/day will be more efficacious than the same dose of iron alone. The specific hypotheses to be tested by the intervention are:

Hypothesis 1: Subjects receiving both iron and vitamin E supplements will have significantly greater changes in serum ferritin (reflecting greater improvement in their iron status), than subjects receiving iron alone after eight weeks of supplementation.

Hypothesis 2: Significantly more subjects receiving both iron and vitamin E supplements will have an improved iron status profile, including ferritin, transferrin saturation, and serum transferrin receptor, than subjects receiving iron alone.

Hypothesis 3 Subjects receiving both iron and vitamin E supplements will have significantly lower levels of inflammatory and oxidant stress biomarkers than subjects receiving iron alone.

Hypothesis 4: (exploratory): The exposure to two months of iron therapy will be associated with significantly altered intestinal bacterial profiles compared to baseline, and at the end of therapy, the placebo group will have a greater predominance of potentially pathogenic bacterial phyla.

ELIGIBILITY:
Inclusion Criteria:

* Between 9-24 months of age
* Weighed 5.5 lbs or more at birth
* Born at 34 week gestation or more

Exclusion Criteria:

* Consumed infant formula within the past 3 months
* Inflammatory bowel disease, cystic fibrosis, liver or kidney disease, cancer, HIV, primary immune deficiencies, anemia unrelated to iron status, chronic blood loss in stool, inherited disorders or iron status, or bleeding or coagulation disorders)
* Previous diagnosis of iron deficiency or iron deficiency anemia
* Previous treatment of iron deficiency or iron deficiency anemia

Ages: 9 Months to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2011-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of iron status, as represented by serum ferritin, to be compared between groups | Up to 8 weeks
  The primary outcome evaluated in this study is iron status, as represented by serum ferritin. Biomarkers include ferritin, hemoglobin, transferrin saturation, and transferrin receptor

SECONDARY OUTCOMES:
Biomarkers of inflammation | Up to 8 weeks
  Secondary outcomes include biomarkers of intestinal and systemic inflammation and of systemic oxidative stress. We will use serum Interleukin (IL)-4, C-Reactive Protein (CRP), and Tumor necrosis factor (TNF)-alpha as indicators of systemic inflammation; and fecal calprotectin as a marker of intestinal (local) inflammation.
Biomarkers of oxidant stress | Up to 8 weeks
  Secondary outcome include biomarkers oxidant stress. We propose to measure urine F2-isoprostanes as a measure of systemic oxidant stress

CONTACTS AND LOCATIONS:
Overall Officials: Nancy F Krebs, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

REFERENCES:
- [Derived] Tang M, Frank DN, Sherlock L, Ir D, Robertson CE, Krebs NF. Effect of Vitamin E With Therapeutic Iron Supplementation on Iron Repletion and Gut Microbiome in US Iron Deficient Infants and Toddlers. J Pediatr Gastroenterol Nutr. 2016 Sep;63(3):379-85. doi: 10.1097/MPG.0000000000001154. PMID 27548249